CLINICAL TRIAL: NCT05835102
Title: Study on the Influence of Nutritional Indices on the Prognosis of Patients With Severe Acute Respiratory Syndrome Coronavirus 2 Infection
Brief Title: Influence of Nutritional Indices on the Prognosis of Patients With SARS-CoV-2 Infection
Status: Recruiting | Type: Observational
Sponsor: Juan Kang (Other)
Responsible Party: Sponsor-Investigator, Juan Kang, associate professor, The Second Affiliated Hospital of Chongqing Medical University
Organization: The Second Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: 2023-19
Record Dates: First submitted 2023-04-23; First posted 2023-04-28 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: COVID-19
Keywords: prognostic nutritional index; geriatric nutritional risk index; pectoralis muscle index; prognosis
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients With SARS-CoV-2 Infection: Patients who test positive for SARS-CoV-2 nucleic acid or SARS-CoV-2 antigen

SUMMARY:
With the decline of virulence after the mutation of the SARS-CoV-2 , based on the national life and health and national development needs, the domestic SARS-CoV-2 infection epidemic prevention policy has changed, and the number of people infected by the SARS-CoV-2 has increased. Nutritional status is an indicator of human health and plays an important role in fighting disease. Malnutrition has been found to correlate with prognosis in patients infected with the SARS-CoV-2 infection . Timely identification and assessment of the patient's nutritional status and early implementation of relevant nutritional intervention are conducive to the recovery of the patient's condition.

In clinical practice, it is necessary to improve nutrition as an aspect of the comprehensive diagnosis and treatment of patients with SARS-CoV-2 infection, but there is still a lack of relevant nutritional indicators or models to simply and accurately assess the nutritional status of patients.The purpose of this study was to evaluate the effects of PNI, NRI, GNRI, albumin level, vitamin D, chest muscle area and density on the clinical characteristics and prognosis of patients with SARS-CoV-2 infection, to find the nutritional predictors of severe disease in patients with SARS-CoV-2 infection, and to establish a simpler and more accurate nutritional evaluation model. To provide evidence for targeted nutritional interventions in patients with SARS-CoV-2 infection.

DETAILED DESCRIPTION:
Patients with SARS-CoV-2 infection attending the Second Affiliated Hospital of Chongqing Medical University were included in the retrospective study. Participants met the inclusion and exclusion criteria. Data to be collected include age, sex, height, and weight at initial treatment; Blood routine, liver function, kidney function, coagulation function, electrolytes, vitamin D, C-reactive protein, ferritin; CT and MRI information; Underlying diseases, complications, treatment options, etc. Follow up patients until discharge or death. After the data collection, statistical methods such as chi-square test and logistic regression analysis were used to evaluate the impact of nutritional factors on the prognosis of patients infected with SARS-CoV-2 infection.

ELIGIBILITY:
Inclusion Criteria:

Patients with a positive SARS-CoV-2 nucleic acid test or a positive SARS-CoV-2 antigen test.

Exclusion Criteria:

1. People with end-stage malignant tumors;
2. Nutritional intake disorders, mainly dependent on enteral and parenteral nutrition supporters;
3. paralyzed;
4. Intravenous drug addicts.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a positive SARS-CoV-2 nucleic acid test or a positive SARS-CoV-2 antigen test.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-12-07 (Estimated); Study Completion 2025-12-09 (Estimated)

PRIMARY OUTCOMES:
Death | October 2022 to January 2023
  Death due to Respiratory failure or other diseases
cure | October 2022 to January 2023
  the patients with SARS-CoV-2 infection are cured and discharged from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Juan Kang, M.D., Study Chair — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No